CLINICAL TRIAL: NCT05788978
Title: Endometriosis Self-Care Behaviors Scale
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 52
Record Dates: First submitted 2023-03-14; First posted 2023-03-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis; Self Care; Behavior; Nursing Role
MeSH Terms: conditions — Endometriosis; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Scale development — Scale development

SUMMARY:
In this study, it was aimed to develop a reliable and valid scale to measure the self-care behaviors of women with endometriosis.

DETAILED DESCRIPTION:
In this study, it was aimed to develop a reliable and valid scale to measure the self-care behaviors of women with endometriosis.This research is of methodological type.Data will be collected by using "Participant Description Questionnaire" and "Self-Care Behaviors Scale in Endometriosis".

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age,
* Diagnosed with endometriosis,
* Having no medical or gynecological problems other than endometriosis,
* Able to read and write,
* Not pregnant,
* No barriers to communication,
* Not diagnosed with a psychiatric illness,
* Volunteer to participate in the study,
* Women who can speak and understand Turkish will be included.
* Followed for at least 6 months,
* Having symptoms related to endometriosis,

Exclusion Criteria:

• Women who incomplete in the data collection forms incompletely will be excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The research will be completed with a minimum of 200 women or a maximum of 420 women diagnosed with endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Self-Care Behaviors Scale in Endometriosis | 9 months
  This scale will be developed to measure the self-care behaviors of women with endometriosis.After the reliability and validity analyzes of the scale, the sub-dimensions of the scale, the number of items and the total score will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamide Arslan Tarus, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No